CLINICAL TRIAL: NCT02144415
Title: A Study to Evaluate the Abuse Potential of EB-1020 Immediate-Release in Healthy Recreational Stimulant Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurovance, Inc. (Industry)
Responsible Party: Sponsor
Organization: Euthymics BioScience, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EB-1020 IR-103
Record Dates: First submitted 2014-05-16; First posted 2014-05-22 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Healthy Volunteers; Drug Users
Keywords: abuse liability; recreational drug user; stimulant; d-amphetamine; ADHD
MeSH Terms: conditions — Drug Misuse; Attention Deficit Disorder with Hyperactivity | interventions — 1-(naphthalen-2-yl)-3-azabicyclo(3.1.0)hexane; Lisdexamfetamine Dimesylate; Dextroamphetamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- EB-1020 400 mg (Experimental): EB-1020 400 mg, administered as four 100-mg IR capsules and 4 matching placebo capsules
  Interventions: Drug: EB-1020 400 mg
- EB-1020 800 mg (Experimental): EB-1020 800 mg, administered as eight 100-mg IR capsules
  Interventions: Drug: EB-1020 800 mg
- lisdexamfetamine 150 mg (Active Comparator): lisdexamfetamine 150 mg, administered as 3 capsules, each containing 1 lisdexamfetamine 50-mg capsule, and 5 matching placebo capsules
  Interventions: Drug: lisdexamfetamine 150 mg
- d-amphetamine 40 mg (Active Comparator): d-amphetamine 40 mg, administered as 4 capsules, each containing two 5-mg d-amphetamine tablets and 4 matching placebo capsules
  Interventions: Drug: d-amphetamine 40 mg
- Placebo (Placebo Comparator): Placebo, administered as 8 matching placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EB-1020 400 mg — 4 x EB-1020 100-mg capsules, and 4 matching placebo capsules
  Arms: EB-1020 400 mg
Drug: EB-1020 800 mg — 8 x EB-1020 100-mg capsules
  Arms: EB-1020 800 mg
Drug: lisdexamfetamine 150 mg — 3 x capsules, each containing 1 lisdexamfetamine 50-mg capsule, and 5 x matching placebo capsules
  Arms: lisdexamfetamine 150 mg
Drug: d-amphetamine 40 mg — 4 x capsules, each containing 2 d-amphetamine 5-mg tablets, and 4 x matching placebo capsules
  Arms: d-amphetamine 40 mg
Drug: Placebo — 8 x matching placebo capsules
  Arms: Placebo

SUMMARY:
This single-center study will be a single-dose, randomized, double-blind, placebo- and active-controlled crossover study with a single inpatient treatment visit. The abuse potential of single oral doses of EB-1020 IR (400 mg, 800 mg) will be compared with that of placebo and d-amphetamine (20 mg, 40 mg; active control) in healthy recreational stimulant users. Subjects will participate in a medical Screening visit (Visit 1), one 4-day inpatient Qualification Phase (Visit 2), one 11-day inpatient Treatment Phase (Visit 3), and a safety Follow-up visit (Visit 4).

DETAILED DESCRIPTION:
Subjects will be randomized to 1 of 10 treatment sequences according to a two 5 x 5 William squares design. To maintain blinding, subjects will be required to ingest eight capsules with approximately 240 mL water on each study drug administration day.

Serial pharmacodynamic (PD) evaluations will be conducted up to 24 hours after each study drug administration. Pharmacokinetic (PK) samples will be obtained to confirm exposure to EB-1020. Safety monitoring will include recording of adverse events (AEs), regular assessments of vital signs measurements, 12-lead electrocardiogram (ECG) findings, and continuous telemetry monitoring for at least 3 hours after study drug administration.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be healthy male nondependent recreational drug users
2. Subjects must be 18 to 55 years old, inclusive.
3. Subjects must have greater than or equal to 10 lifetime nontherapeutic experiences with central nervous system (CNS) stimulants (e.g., amphetamines, cocaine, methylphenidate), greater than or equal to 1 nontherapeutic use of prescription stimulants within the 12 months prior to Screening, and greater than or equal to 1 nontherapeutic use of a CNS stimulant within the 12 weeks prior to Screening.

Exclusion Criteria:

1. Subjects that are deemed medically unsuitable or unlikely to comply with the study protocol for any reason.
2. Subjects who do not pass Qualification Phase criteria to be eligible for the Treatment Phase.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Maximum effect (Emax) on Drug Liking visual analog scale (VAS) | within 24 hours post-dose
  Drug liking VAS is one of the measures of balance of effects that assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 millimeter (mm) bipolar visual analogue scale (VAS) anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), on the left with "strong disliking" (score of 0 mm) and on the right with "strong liking" (score of 100 mm).

SECONDARY OUTCOMES:
Drug Liking VAS (minimum effect [Emin] and time-averaged area under the effect curve to 12 hours after study drug administration [TA_AUE]) | within 24 hours post-dose
  Drug liking VAS is one of the measures of balance of effects that assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 millimeter (mm) bipolar visual analogue scale (VAS) anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), on the left with "strong disliking" (score of 0 mm) and on the right with "strong liking" (score of 100 mm).
Overall Drug Liking VAS (Emax/Emin) | within 24 hours post-dose
  Overall drug liking VAS is one of the measures of balance of effects that assesses the participant's global perception of drug liking (that is, effects over the whole course of the drug experience including any carryover effects). A 100 mm bipolar VAS is used to assess response based on a score ranging from 0 mm to 100 mm (0 mm = "strong disliking", 50 mm= "neither like nor dislike", and 100 mm= "strong liking").
Take Drug Again VAS (Emax) | within 24 hours post-dose
  Take drug again VAS is one of the measures of balance of effects. It is a subjective assessment of the degree to which a participant would desire to take the drug again if given the opportunity. It is presented on a 100 mm bipolar VAS with score ranging from 0 mm to 100 mm (score of 0 mm = "definitely not", 50 mm = "do not care", and 100 mm = "definitely so").
High VAS (Emax and TA_AUE) | within 24 hours post-dose
  High VAS is one of the measures of positive effects that assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm= definitely not) to 'extremely' (score of 100 = definitely so).
Good Effects VAS (Emax and TA_AUE) | within 24 hours post-dose
  Good drug effects VAS is one of the measures of positive effects that assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm= definitely not) to 'extremely' (score of 100 mm= definitely so).
Bad Effects VAS (Emax and TA_AUE) | within 24 hours post-dose
  Bad effects VAS is one of the measures of negative effects that assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm= definitely not) to 'extremely' (score of 100 mm= definitely so).
Nausea VAS (Emax and TA_AUE) | within 24 hours post-dose
  Nausea VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm).
ARCI-A scale (Emax and TA_AUE) | within 24 hours post-dose
  ARCI-A is measure of other stimulant effects. It is a set of 13 questions in which each question contributes to total score. Participants select 'False' / 'True' for response. One point given for each response that agrees with scoring direction, true items receive score of 1 if answer 'True', false items receive score of 1 if answer 'False'. No points if answer is opposite to scoring direction. Score range: 0 to 13, higher score indicated higher other subjective effects.
ARCI-BG scale (Emax and TA_AUE) | within 24 hours post-dose
  ARCI-BG is measure of other subjective effects. It is a set of 13 questions in which each question contributes to total score. Participants select 'False' / 'True' for response. One point given for each response that agrees with scoring direction, true items receive score of 1 if answer 'True', false items receive score of 1 if answer 'False'. No points if answer is opposite to scoring direction. Score range: 0 to 13, higher score indicated higher other subjective effects.
Alertness/Drowsiness VAS (Emax and TA_AUE) | within 24 hours post-dose
  Alertness/Drowsiness VAS is one of the measures of sedative effects. It is scored using a 100 mm bipolar VAS anchored in the center with a neutral anchor of "neither drowsy nor alert" (score of 50 mm), on the left with "very drowsy" (score of 0 mm) and on the right with "very alert" (score of 100 mm).
Agitation/Relaxation VAS (Emax and TA_AUE) | within 24 hours post-dose
  Agitation/Relaxation VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm).
Any Effects VAS (Emax and TA_AUE) | within 24 hours post-dose
  Any drug effects VAS is one of the measures of other subjective effects. It assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm= definitely not) to 'extremely' (score of 100 mm= definitely so).
Drug Similarity VAS (score at 12 hours after study drug administration) | within 24 hours post-dose
  Drug similarity VAS is one of the measures of other subjective effects. It assesses the similarity of the drug recently received by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm= not at all similar) to 'extremely' (score of 100 mm= very similar). Recently received drugs were compared with placebo, benzodiazepines, codeine/morphine, Tetrahydrocannabinol (THC), pseudoephedrine.
Safety and tolerability of EB-1020 as assessed by AEs | Up to 6 weeks
Safety and tolerability of EB-1020 by laboratory assessments | Up to 6 weeks
Safety and tolerability of EB-1020 as assessed by 12-lead ECGs | Up to 6 weeks
Safety and tolerability of EB-1020 as assessed by vital signs | Up to 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Vince and Associates Clinical Research, Inc., Overland Park, Kansas, United States